CLINICAL TRIAL: NCT02575599
Title: Assessment of a Web-based Guided Self-Determination Intervention for Adults With Type 2 Diabetes in General Practice
Brief Title: Web-based Guided Self-Determination Intervention for Adults With Type 2 Diabetes in General Practice
Acronym: DiaWeb
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Stavanger (Other)
Collaborators: Bergen University College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DIW 221065
Record Dates: First submitted 2015-10-09; First posted 2015-10-14 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2016-11

CONDITIONS: Type 2 Diabetes
Keywords: Self-management; web-based; quantitative approach
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle counselling (Active Comparator): Intervention group: Eighty six adults with type 2 diabetes will be recruited from the general practices where the trained nurses in Guided self-determination programme are working.
  Interventions: Behavioral: Guided self-determination programme (GSD)
- Regular consultation (No Intervention): Control group: Eighty six adults with type 2 diabetes will be recruited from general practices with employed registered nurses without the Guided self-determination training.

INTERVENTIONS:
Behavioral: Guided self-determination programme (GSD) — The GSD intervention consist of four e-consultations with structured reflection sheets. Reflection sheets are intended to increase patients' ability to express their views and prepare them for active participation in the care process. Through the web-based platform, the subsequent four e-consultations will allow for communication between patients and nurses. The platform allows the participants to fill in the reflection sheets using their own words and drawings to express their own experiences with self-management as well as to formulate behavioral goals and plans to achieve their goals. It also permits feedback from the nurses on these reflections sheets via secure emails. Each person will be able to access the web-based program from his or her own computers or other electronic devices.
  Arms: Lifestyle counselling

SUMMARY:
The overall aim of this study is to assess the effectiveness of a web-based Guided Self-Determination program among adults with type 2 diabetes in general practice in order to improve diabetes self-management behaviours and HbA1c through enhanced patient activation, self-care competence, and autonomy.

DETAILED DESCRIPTION:
Web-based self-management programs have the potential to support adults with type 2 diabetes in managing their disease condition. However, improving health care outcomes through self-management interventions have shown somewhat ambiguous results. Therefore, it is suggested that interventions should be theory-based and incorporate well-defined counselling methods and techniques for behavioural change. To meet these challenges, the overall aim of this study is to assess the effectiveness of a theory-driven web-based Guided Self-Determination intervention among adults with type 2 diabetes in general practice in order to enable adults with diabetes to use their individual resources to self-manage their condition and reach treatment goals.

A complex intervention design based on the framework of UK Medical Research Council is employed as a guide for developing and evaluating the intervention.

This study consists of three phases:

1. the modelling phase adapting the original Guided Self-Determination program to adults with type 2 diabetes, using a qualitative design
2. feasibility assessment of the adapted intervention on the web, employing qualitative and quantitative methods and
3. evaluating the effectiveness of the intervention on diabetes self-management behaviours and HbA1c, using a quasi-experimental design.

The two first phases will provide important information about the development of the intervention and its acceptability, whereas the third phase will assess the effect on health care outcomes of this systematically developed intervention.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes of duration ≥ 3 months
* Ability to communicate in Norwegian
* Access to the internet and bank ID

Exclusion Criteria:

* Patients with cognitive impairment
* Patients with severe co-morbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
The Patient Activation Measure (PAM) | Assessing change between three time points: Change from baseline at 12-16 weeks, and change from 12- 16 weeks at 6 months

SECONDARY OUTCOMES:
The Health Care Climate Questionnaire (HCCQ) | Assessing change between three time points: Change from baseline at 12- 16 weeks, and change from 12- 16 weeks at 6 months
Perceived Competence for Diabetes Scale (PCDS) | Assessing change between three time points: Change from baseline at 12- 16 weeks, and change from 12- 16 weeks at 6 months
Treatment Self-Regulation (TSRQ) | At three time points: at baseline, 12-16 weeks later at the end of the intervention and six months after finishing the intervention.
Diabetes Management Self-efficacy Scale (SE-type 2 diabetes) | Assessing change between three time points: Change from baseline at 12-16 weeks, and change from 12-16 weeks at 6 months
Summary of diabetes self-care activities (SDSCA) | Assessing change between three time points: Change from baseline at 12-16 weeks, and change from 12-16 weeks at 6 months
The WHO 5-item Well-Being Index (WHO-5) | Assessing change between three time points: Change from baseline at 12-16 weeks, and change from 12-16 weeks at 6 months
Diabetes Distress Scale (DDS) | Assessing change between three time points: Change from baseline at 12-16 weeks, and change from 12- 16 weeks at 6 months
Glycosylated haemoglobin (HbA1c) | Assessing change between three time points: Change from baseline at 12-16 weeks, and change from 12-16 weeks at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marit Graue, Professor, Study Director — Bergen University College, Inndalsveien 28, 5063 Bergen, Norway

REFERENCES:
- [Derived] Karlsen B, Oftedal B, Stangeland Lie S, Rokne B, Peyrot M, Zoffmann V, Graue M. Assessment of a web-based Guided Self-Determination intervention for adults with type 2 diabetes in general practice: a study protocol. BMJ Open. 2016 Dec 13;6(12):e013026. doi: 10.1136/bmjopen-2016-013026. PMID 27965253